CLINICAL TRIAL: NCT03977220
Title: Phase I Study: Nab-paclitaxel Combined With S-1 Treating Diffuse Type of Stage Ⅲ Gastric Cancer as Adjuvant Setting (NORDICA)
Brief Title: Nab-paclitaxel Combined With S-1 Treating Diffuse Type of Stage Ⅲ Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Chairman for the department of oncology, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NORDICA
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel combined with S-1 (Experimental): Nab-paclitaxel combined with S-1 treating diffuse type of stage Ⅲ gastric cancer as adjuvant setting
  Interventions: Drug: Nab-paclitaxel combined with S-1

INTERVENTIONS:
Drug: Nab-paclitaxel combined with S-1 — Nab-paclitaxel combined with S-1 treating diffuse type of stage Ⅲ gastric cancer as adjuvant setting

SUMMARY:
Investigators assessed the effectiveness of Nab-paclitaxel combined with S-1 treating diffuse type of stage Ⅲ gastric cancer as adjuvant setting

DETAILED DESCRIPTION:
Adjuvant chemotherapy is still the standard of care for stage Ⅲ gastric cancer. Till now, oxaliplatin with capecitabine or S1 still the standard chemotherapy regimen. Howerver, the prognosis of diffuse type gastric cancer patients is still poor even after adjuvant chemotherapy of XELOX or S1 regimen. Several retrospective, single institutional studies have shown that the addition of Nab-paclitaxel to S1 can prolong the survival of advanced gastric cancer with diffuse type.However, the effection of Nab-paclitaxel and S1 is unknown in diffuse gastric cancer patients after radical surgery. We assessed the effectiveness of radical surgery following docetaxel, nab-pacitaxel and S1 therapy for gastric cancer with diffuse type.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer patients after radical resection
* diffuse type gastric cancer stage III

Exclusion Criteria:

* Patients who have metastasis disease
* Patients who can not tolerate chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended dose for Phase II study | through study completion, an average of 2 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui Y, Yu Y, Yu S, Li W, Wang Y, Li Q, Liu T. Phase I study of adjuvant chemotherapy with nab-paclitaxel and S-1 for stage III Lauren's diffuse-type gastric cancer after D2 resection (NORDICA study). Cancer Med. 2023 Jan;12(2):1114-1121. doi: 10.1002/cam4.4966. Epub 2022 Jun 25. PMID 35751496